CLINICAL TRIAL: NCT06787430
Title: Evaluating the Effects of Nicorandil on Microvascular Dysfunction in Patients With ST-segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Effects of Nicorandil on Microvascular Dysfunction in Patients With STEMI Undergoing Primary PCI
Acronym: NORMAL
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-2375
Record Dates: First submitted 2024-12-26; First posted 2025-01-22 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: STEMI - ST-segment Elevation Myocardial Infarction
Keywords: Nicorandil; STEMI; microvascular dysfunction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Nicorandil; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nicorandil group (Experimental): In the nicorandil group, intracoronary nicorandil 3mg dissolved in 3ml saline was given within 30 seconds at two time points, one was when the guidewire or ballon passed the lesion and the blood flow was regained, and another was the time before the stent was implanted.
  Interventions: Drug: nicorandil
- Control group (Placebo Comparator): In the control group, 3ml saline was given within 30 seconds at the same time points in nicorandil group.
  Interventions: Drug: Saline (NaCl 0,9 %) (placebo)

INTERVENTIONS:
Drug: nicorandil — In the nicorandil group, intracoronary nicorandil 3mg dissolved in 3ml saline was given within 30 seconds at two time points, one was when the guidewire or ballon passed the lesion and the blood flow was regained, and another was the time before the stent was implanted.
  Arms: Nicorandil group
Drug: Saline (NaCl 0,9 %) (placebo) — In the control group, 3ml saline was given intracoronary through the guiding catheter within 30 seconds at the same time points in nicorandil group.
  Arms: Control group

SUMMARY:
Despite the success of restoration of epicardial blood flow by the primary percutaneous coronary intervention (PPCI), approximately one half of patients with ST-segment elevation myocardial infarction (STEMI) have failed myocardial reperfusion, namely microvascular dysfunction. Previous studies have shown that coronary microvascular damage significantly impacts the prognosis of patients with STEMI. Therefore, restoration of microvascular function is quite important during the PPCI procedures. Recent clinical trials found that nicorandil, a hybrid ATP-sensitive potassium channel opening agent, improved microvascular function, prevented no-reflow phenomenon, and had beneficial cardioprotective effects in patients receiving PPCI. However, there was a lack of evidence on the protective effects of nicorandil on microvascular function. The coronary angiography-derived IMR (AMR) is a novel wire-free technology developed for fast computation of IMR in patients undergoing coronary angiography, thereby enabling the quantification of coronary microcirculation of patients. This study is aimed to investigate the effects of nicorandil on microvascular dysfunction as evaluated by AMR in patients with STEMI.

DETAILED DESCRIPTION:
This study is aimed to investigate the effects of nicorandil on microvascular dysfunction as evaluated by AMR in patients with STEMI.

This study is a prospective, single-center, double-blind, randomized controlled study, evaluate the effects of nicorandil on nicorandil on microvascular dysfunction in patients with STEMI undergoing primary PCI.

The inclusion criteria are as following: Age between 18-80; Diagnosis of STEMI and indicating for primary PCI; Diagnostic coronary angiography showed definite culprit vessel and primary PCI was planned to treat the culprit vessel; Reference vessel diameter of culprit vessel was greater than 2.0 mm; There was no flow-limiting stenosis for the non-culprit vessels; Understand the aim of this trial and agree to sign the informed consent form.

The exclusion criteria are as following: Acute in- stent thrombosis or in-stent stenosis lesions of culprit vessel; Balloon angioplasty rather than stent was planned for the culprit vessel; Allergic to nicorandil or systolic arterial pressure was less than 85mmHg before procedure; Vessel with twisted shape that was unable to be measured using AMR; Oral or intravenous use of nicorandil within one month; Cardiac shock needing mechanical support; Severely hepatic dysfunction; Severely renal failure needing hemodialysis; Contraindicated for coronary angiography or primary PCI; Culprit vessels of left main or graft vessels; Pregnant or nursing; Others that investigators think should excluded.

Patients were randomized into nicorandil group and control group with ratio of 1:1. In the nicorandil group, intracoronary nicorandil 3mg dissolved in 3ml saline was given within 30 seconds at two time points, one was when the guidewire or ballon passed the lesion and the blood flow was regained, and another was the time before the stent was implanted. In the control group, 3ml saline was given intracoronary through the guiding catheter within 30 seconds at the same time points in nicorandil group. All the procedure details including strategies, decision of intravascular imaging, other medications during procedures were decided by operators.

The angiography-derived microcirculatory resistance (AMR) is a wire-free and adenosine-free index, which aims at providing a valid alternative to invasive wire-based IMR assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80
* Diagnosis of STEMI and indicating for primary PCI
* Diagnostic coronary angiography showed definite culprit vessel and primary PCI was planned to treat the culprit vessel.
* Reference vessel diameter of culprit vessel was greater than 2.0 mm
* There was no flow-limiting stenosis for the non-culprit vessels.
* Understand the aim of this trial and agree to sign the informed consent form.

Exclusion Criteria:

* Acute in- stent thrombosis or in-stent stenosis lesions of culprit vessel.
* Balloon angioplasty rather than stent was planned for the culprit vessel.
* Allergic to nicorandil or systolic arterial pressure was less than 85mmHg before procedure
* Vessel with twisted shape that was unable to be measured using AMR
* Oral or intravenous use of nicorandil within one month.
* Cardiac shock needing mechanical support.
* Severely hepatic dysfunction.
* Severely renal failure needing hemodialysis.
* Contraindicated for coronary angiography or primary PCI.
* Culprit vessels of left main or graft vessels.
* Pregnant or nursing.
* Others that investigators think should excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The value of post-PCI AMR | The time immediate after primary PCI
  AMR was obtained by analyzing the last angiography video of culprit vessel after procedure. AMR was analyzed by sophisticated technicians who were unaware of the group division.

SECONDARY OUTCOMES:
Prevalence of slow flow or no-flow during procedure | During primary PCI procedure
ST-segment resolution two hours after primary PCI | Two hours after primary PCI
  Analyze the elevated leads of EKG two hours after primary PCI
In-hospital peak troponin level | From the enrollment to 7 days after primary PCI
Prevalence of hypotension during procedure | During primary PCI procedure
  Prevalence of hypotension during procedure: defined by systolic arterial pressure less than 85mmHg or systolic arterial pressure dropped greater than 40mmHg after the use of nicorandil and lasted for 15 minutes.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang X, Guo Q, Guo R, Guo Y, Yan Y, Gong W, Zheng W, Wang H, Ai H, Que B, Xu L, Huo Y, Fearon WF, Nie S. Coronary angiography-derived index of microcirculatory resistance and evolution of infarct pathology after ST-segment-elevation myocardial infarction. Eur Heart J Cardiovasc Imaging. 2023 Nov 23;24(12):1640-1652. doi: 10.1093/ehjci/jead141. PMID 37319341
- [Background] Hirohata A, Yamamoto K, Hirose E, Kobayashi Y, Takafuji H, Sano F, Matsumoto K, Ohara M, Yoshioka R, Takinami H, Ohe T. Nicorandil prevents microvascular dysfunction resulting from PCI in patients with stable angina pectoris: a randomised study. EuroIntervention. 2014 Jan 22;9(9):1050-6. doi: 10.4244/EIJV9I9A178. PMID 24457276
- [Background] Qian G, Zhang Y, Dong W, Jiang ZC, Li T, Cheng LQ, Zou YT, Jiang XS, Zhou H, A X, Li P, Chen ML, Su X, Tian JW, Shi B, Li ZZ, Wu YQ, Li YJ, Chen YD. Effects of Nicorandil Administration on Infarct Size in Patients With ST-Segment-Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention: The CHANGE Trial. J Am Heart Assoc. 2022 Sep 20;11(18):e026232. doi: 10.1161/JAHA.122.026232. Epub 2022 Sep 8. PMID 36073634